CLINICAL TRIAL: NCT06276595
Title: Telling Our Daughters Our Story: Pre-Conception Health Program for American Indian Girls as They Transition to Adulthood
Brief Title: Telling Our Daughters Our Story
Acronym: TODOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: White Mountain Apache Tribe (Unknown); Native American Research Center for Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB00009466
Record Dates: First submitted 2024-02-16; First posted 2024-02-26 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Substance Use; Sexual Behavior
MeSH Terms: conditions — Substance-Related Disorders; Sexual Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TODOS Intervention (Experimental): Participants in the TODOS Intervention Group will receive the intervention "Nowhi Isdza bit Nadagoldi": Telling Our Daughters Our Story. They will receive 11 intervention sessions of 60-90 minutes over 11 weeks.
  Interventions: Behavioral: Nowhi Isdza bit Nadagoldi: Telling Our Daughters Our Story (TODOS)
- Control condition - 3 Monthly Group Activities in the Community (Other): Children and their female caregivers randomized to the control group will receive 3 group sessions delivered monthly for three months. The first group session will occur at a community center and will consist of a meal and ice breaker activities. The second group session will consist of going to a movie at the local movie theatre. The third group session will consist of going bowling at the local bowling alley.
  Interventions: Behavioral: Control condition - 3 Monthly Group Activities in the Community

INTERVENTIONS:
Behavioral: Nowhi Isdza bit Nadagoldi: Telling Our Daughters Our Story (TODOS) — The TODOS program consists of 11 weekly sessions conducted with girls ages 8-11 and their female caregivers. Five of the 11 sessions will be taught to small groups, and 6 of the Each of the sessions (group and individual) will be 60-90 minutes in duration and delivered by a trained Family Health Coach (FHC). Group sessions will take place at a local community center in a private room.
  Arms: TODOS Intervention
Behavioral: Control condition - 3 Monthly Group Activities in the Community — The control condition consists of 3 group sessions delivered monthly for three months. The first group session will occur at a community center and will consist of a meal and ice breaker activities. The second group session will consist of going to a movie at the local movie theatre The third group session will consist of going bowling at the local bowling alley.
  Arms: Control condition - 3 Monthly Group Activities in the Community

SUMMARY:
The objective of this research study is to evaluate a culturally grounded program among American Indian (AI) female children and the children's female caregivers. This project will evaluate the impact of "Nowhi Isdza bit Nadagoldi: Telling Our Daughters Our Story (henceforth referred to as TODOS) on associated risk and protective factors for early substance use and sexual debut through a randomized controlled trial on the White Mountain Apache (WMA) reservation. The investigators will examine whether the TODOS program effectively reduces risk factors and improves protective factors associated with early substance use and sexual debut, with long term goals of reducing teen pregnancy and teen substance use.

DETAILED DESCRIPTION:
The investigators will employ a randomized controlled trial (RCT) design to assess the preliminary impact of the TODOS program on many factors, including improving cultural knowledge, family engagement in Apache culture, mother daughter communication, self-esteem, self-efficacy, social support, attitudes about risky behaviors, and knowledge of reproductive health and substance use. Participants will be caregivers of girls ages 8-11 years.

The TODOS program consists of 11 weekly sessions conducted with girls ages 8-11 and the girl's female caregivers. Five of the 11 sessions will be taught to small groups of girls and the girl's mothers, and 6 of the sessions will be taught to individual girl/female caregivers' dyads. The choice to use a mix of group- and home-based sessions is based on findings from the formative phase about preference that certain topics be taught in groups, and certain topics be taught in individual dyads. Each of the sessions (group and individual) will be 60-90 minutes in duration and delivered by a trained Family Health Coach (FHC).

The investigators will enroll up to 94 dyads into four cohorts, each consisting of 18-26 dyads. Dyads will receive either the TODOS program or a control condition. The control condition will consist of 3 group sessions delivered monthly for three months. The investigators will evaluate the TODOS program's feasibility through process data including attendance forms and session summary feedback forms completed by the FHCs. The investigators will assess program acceptability immediately after program completion through implementation assessments completed by caregiver and children participants. The investigators will assess the program's impact on key outcomes immediately after program implementation, 6-month and 12-month post program implementation.

ELIGIBILITY:
Inclusion Criteria for Caregivers:

* Female > 18 years of age
* Self-identify as Apache
* Be a caregiver of a girl 8-11 years old who is available to enroll in the study
* Living within 50 miles of the Whiteriver or Fort Apache, Arizona Johns Hopkins program offices
* Willing to complete all implementation and follow-up assessments
* Willing to be randomized
* Speaks and reads English

Inclusion Criteria for Child Participants:

* Female, 8-11 years old
* Have a caregiver enrolled in the study
* Living within 50 miles of the Whiteriver or Fort Apache, Arizona Johns Hopkins program offices
* Willing to be randomized
* Willing to complete all implementation and follow-up assessments
* Speaks and reads English
* Not cognitively or visually impaired (able to complete questionnaires)

Exclusion Criteria:

* Inability to participate in full intervention or evaluation (e.g., planned move, residential treatment, cognitive impairment, etc.)

Min Age: 8 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — This is a program for female caregivers of female children.
Enrollment: 183 (Actual)
Dates: Start 2019-03-30 (Actual); Primary Completion 2022-03-22 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
Change in child cultural knowledge score on knowledge assessment | Baseline, 11 weeks, 6 months, 12 months
  Using a questionnaire developed by the study team, investigators will measure change in knowledge from baseline to immediately following the intervention and 6 months and 12 months after program completion via a knowledge assessment completed by the child. This is a 4- question assessment that is on a 5-point Likert scale (score: 0-20) A higher score indicates higher (greater) knowledge.
Change in average score on risky behaviors assessment | Baseline, 11 weeks, 6 months, 12 months
  Using a questionnaire developed by the study team, the investigators will assess the impact of the TODOS program on child attitudes related to risky behaviors via a 6-item assessment on a 5-point Likert scale (score: 0-30). Investigators will measure change in knowledge from baseline to immediately following the intervention and 6 months and 12 months after program completion via a knowledge assessment completed by the child. A higher score indicates better attitudes (less endorsement of) risk behaviors.
Change in child reproductive health knowledge via a reproductive health knowledge questionnaire | Baseline, 11 weeks, 6 months, 12 months
  Using a questionnaire developed by the study team, investigators will measure change in knowledge from baseline to immediately following the intervention and 6 months and 12 months after program completion via a 3-question knowledge assessment completed by the child (score 0-100). A higher score indicates more knowledge.

CONTACTS AND LOCATIONS:
Overall Officials: Mary Barlow, PhD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- White Mountain Apache Center for Indigenous Health, Whiteriver, Arizona, United States

IPD SHARING:
Plan to Share IPD: No